CLINICAL TRIAL: NCT05000476
Title: Effect of Eye Mask and Earplugs on Prevention of Delirium in Intensive Care Patients
Brief Title: Using Eye Mask and Earplugs on Prevention of Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Gülşen Kılıç, Nurse, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GulsenK
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Delirium
Keywords: Delirium; Intensive care unit; Earplugs; Eyemask; Nursing
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nurse Education and Environmental Regulation (Other): Clinical nurses will be given training on delirium risks, diagnosis, prevention and management. In order to implement the interventions, environmental arrangements will be made in the intensive care units in the light of the training given, and the nurses will record which attempts are made during the day with the daily follow-up form.
  Interventions: Other: Nurse Education and Environmental Regulation
- Eye mask and earplugs (Experimental): Patients will be monitored for 3 days starting from their hospitalization.
  Along with the regulations, each patient will be assisted by the intensive care nurses for 3 days between 23:00 p.m. - 06:00 a.m. for the use of eye mask and earplugs.
  Interventions: Other: eye mask and earplugs
- Control (No Intervention): With the adjustments made, theywill receive the usual care for 3 days.

INTERVENTIONS:
Other: eye mask and earplugs — Materials similar to those offered on long commercial flights
  Arms: Eye mask and earplugs
Other: Nurse Education and Environmental Regulation — providing orientation to the patient (frequent orientation of the patient to the place, time and person), cognitive stimulation (objects such as clocks and calendars in the patient's field of view), reducing noise and light (minimizing monitors and fluid infusion pump alarms at night), providing early mobilization ( passive-active joint movements, sitting and walking in bed), reducing social deprivation (receiving visitors, telephone calls)
  Arms: Nurse Education and Environmental Regulation

SUMMARY:
This research is planned as a randomized controlled experimental study to examine the effect of using eye mask and earplugs in preventing delirium with evidence-based nonpharmacological nursing interventions in intensive care units.

DETAILED DESCRIPTION:
In the prevention of delirium, the necessity of using a multicomponent, nonpharmacological interventions is emphasized and focused on nursing interventions. In this regard, it is believed that the use of eye mask and ear plugs, which have recently started to take place in the guides, as well as known evidence-based nursing interventions, will provide nurses with power to improve delirium-related outcomes.

The research is expected to consist of intervention and control groups older than 18, volunteering to participate in the research, which the expected length of stay in the ICU more than 24 hours at Başkent University Ankara Hospital. Data will be collected through Patient Information Form, APACHE II, Glasgow Coma Scale, Richmond Sedation Agitation Scale, Nursing-Delirium Screening Scale, Richard-Campbell Sleep Scale and Daily Monitoring Form. In preparation step of the research, nurses will be trained, guidelines are required for nurses, necessary interventions will be planned. At the application stage , after determining the experimental and control groups, eye mask and ear plugs will be given before going to sleep in addition to the patients in the experimental group, before going to sleep, and followed for three days. Also, it will be examined through a semi-structured interview technique for the examination of patients in the experimental group.It is believed that the early diagnosis of delirium, nonpharmacological interventions to be implemented will affect the diagnosis-treatment costs positively by reducing morbidity and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* The expected duration of stay in the intensive care unit is more than 24 hours.
* In the first 24 hours of hospitalization,
* On mechanical ventilation, conscious patients
* Patients who volunteered to participate in the study
* Not using sleeping pills* * Prescription drugs (benzodiazepines, nonbenzodiazepines), quetiapine, antihistamines, antidepressants used for their sedative effects

Exclusion Criteria:

* illness
* Suspected or approved drug or alcohol poisoning
* Contraindication to the use of earplugs or eye masks (eg facial trauma or other safety concerns)
* Patients using hearing aids
* Severe neurological deficits defined as coma (Richmond Agitation Sedation Score <-4 or -5 (deeply sedated and coma) due to cranial trauma, malignancy, anoxic brain injury, or cerebral edema)
* Having a known cognitive disorder (such as dementia, Alzheimer's, psychosis.)
* Patients with a Glasgow coma scale (GCS) of 8 and below

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-09-21 (Estimated)

PRIMARY OUTCOMES:
delirium | three days
  The effect of non-pharmacological interventions on the prevalence of delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)